CLINICAL TRIAL: NCT06937567
Title: Exploratory Study on the Safety and Preliminary Efficacy of UCLH80-1 Cells in Patients With CDH17-Positive Advanced Malignant Solid Tumors
Brief Title: CDH17 CAR-T Therapy in Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Weijia Fang, MD, Chief doctor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLH801-II
Record Dates: First submitted 2024-12-24; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer; Colorectal Carcinoma; Gastric Cancer, Metastatic; Pancreatic Adenocarcinoma (Ductal Adenocarcinoma); Multiple Cancer
Keywords: CAR-T; CDH17
MeSH Terms: conditions — Biliary Tract Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CDH17 CAR-T treatment arm (Experimental): In this study, patients with advanced malignant solid tumors with positive CDH17 expression will be enrolled in a traditional "3+3 design" dose climb test.
  The initial dose of cell therapy in this clinical study was set at 1.0×106/Kg and the maximum dose was set at 6.0×106/Kg.
  Interventions: Biological: CDH17 CAR-T

INTERVENTIONS:
Biological: CDH17 CAR-T — The initial dose of cell therapy in this clinical study was set at 1.0×106/Kg and the maximum dose was set at 6.0×106/Kg.

SUMMARY:
The investigational product used in this study, UCLH801 cells, is a CAR-T cell therapy specifically targeting CDH17. The proposed indication includes CDH17-positive advanced solid tumors, such as but not limited to colorectal cancer, gastric cancer, pancreatic cancer, biliary tract tumors, neuroendocrine tumors, ovarian cancer, and lung cancer. The primary objective of this study is to evaluate the safety and tolerability of UCLH801 cells in patients with CDH17-positive advanced malignant solid tumors. The secondary objectives include assessing the preliminary efficacy of UCLH801 cells, their pharmacokinetics and pharmacodynamics in the body, and their immunogenicity.

This study aims to observe how the infusion of UCLH801 cells affects patients 's body, including any discomfort or changes in laboratory test results. Additionally, it will evaluate whether UCLH801 cells have any effect on tumor. Furthermore, the study will investigate how UCLH801 cells are metabolized; the mechanisms through which they exert their effects, and how to develops any immune response or rejection against UCLH801 cells.

DETAILED DESCRIPTION:
The trial progresses through sequential Phase Ia (dose-finding) and Phase Ib (dose-expansion) stages. Phase Ia cessation triggers include either confirmation of Recommended Phase II Dose (RP2D) or investigator-verified favorable therapeutic index at any dose level. Post-Phase Ia completion, protocol amendment submission to the Institutional Review Board precedes Phase Ib initiation, featuring multi-cohort expansion (n=9-18/cohort) across specified malignancies: colorectal adenocarcinoma (CRC), gastric carcinoma (GC), high-grade serous ovarian carcinoma (HGSOC), breast cancer (BC), non-small cell lung cancer (NSCLC), SCLC, metastatic castration-resistant prostate cancer (mCRPC), clear cell renal cell carcinoma (ccRCC), and cervical squamous cell carcinoma (CSCC), etc.

This study has 3 dose levels and follows a "3+3 design," with an estimated enrollment of 9 to 18 subjects. The final sample size will depend on the occurrence of dose-limiting toxicities (DLTs), the number of dose escalation groups before observing DLTs, and the maximum tolerated dose (MTD). Considering the possibility of cell production preparation failure or other reasons (such as rapid disease progression during cell preparation) leading to subjects ultimately being unable to receive cell infusion therapy, the number of participants in the cell collection and preparation process may be greater than the planned number of cases.

The observation period for dose-limiting toxicity (DLT) is set from the start of cell infusion to 4 weeks after the completion of cell infusion (D0 to D28).

The starting dose of cell infusion therapy in this clinical study is set at 1.0×10^6/Kg, and the maximum dose is set at 6.0×10^6/Kg.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed malignant solid tumors, including but not limited to colorectal cancer, gastric cancer, pancreatic cancer, and biliary tract tumors.
* Patients must have failed standard treatments, be intolerant to standard treatments, or lack effective treatment options.
* At least one measurable lesion as defined by RECIST v1.1 criteria.
* Tumor tissue must be available either from prior tumor biopsy or by providing new tumor specimens.
* Tumor specimens must be confirmed as CDH17-positive by immunohistochemistry (IHC) or immunocytochemistry (ICC) staining.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival time ≥ 3 months.
* Appropriate organ function: hematological: Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Absolute lymphocyte count (ALC) ≥ 0.5 × 10⁹/L. Hemoglobin (HGB) ≥ 80 g/L; Platelet count (PLT) ≥ 75 × 10⁹/L. Liver Function: aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0 × ULN (≤ 5.0 × ULN for patients with primary liver tumors or liver metastases); total bilirubin ≤ 1.5 × ULN (≤ 3.0 × ULN for patients with primary liver tumors or liver metastases; ≤ 3 × ULN for Gilbert's syndrome with direct bilirubin ≤ 1.5 × ULN). Coagulation: international normalized ratio (INR) ≤ 1.5 × ULN (unless on therapeutic anticoagulants); activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (unless on therapeutic anticoagulants). Renal Function: serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 mL/min (based on Cockcroft-Gault formula). Cardiac Function: left ventricular ejection fraction (LVEF) ≥ 50% (confirmed by echocardiography). Pulmonary Function: resting oxygen saturation (SpO₂) > 92% without supplemental oxygen.
* Female participants of childbearing potential must have a negative pregnancy test.
* Female participants of childbearing potential or male participants with partners of childbearing potential must agree to use effective contraception during the study and for 1 year after the final cell infusion.
* Willingness to sign the informed consent form, demonstrating understanding of the study and agreement to comply with study procedures.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Positive hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) with peripheral HBV DNA levels above the lower limit of detection.
* Positive hepatitis C virus (HCV) antibody with peripheral HCV RNA levels above the lower limit of detection.
* Positive HIV antibody.
* Positive syphilis-specific and non-specific antibody tests.
* Non-hematological toxicity from prior treatment (surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) has not resolved to ≤ CTCAE grade 1 (except for hair loss and peripheral sensory neuropathy).
* Prior allogeneic tissue or organ transplant (including bone marrow, stem cell, liver, kidney, etc.), except for transplants not requiring immunosuppression (e.g., corneal or hair transplantation).
* Patients who have previously received CDH17 CAR-T therapy, except those who received CAR-T infusion within this study.
* Underwent major surgery within 4 weeks prior to signing informed consent and has not fully recovered, or has a history of serious unresolved trauma.
* Known central nervous system (CNS) metastases (with exceptions for asymptomatic brain metastases or stable clinical symptoms).
* Severe active infections or pulmonary diseases requiring systemic corticosteroid treatment within 6 months prior to signing informed consent.
* Symptomatic congestive heart failure (NYHA class II-IV), severe aortic stenosis, or symptomatic mitral stenosis.
* ECG showing QTc > 450 ms or QTc > 480 ms with bundle branch block.
* Uncontrolled hypertension (SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg).
* Cerebrovascular accidents within 6 months prior to signing informed consent.
* Active, chronic, or recurrent severe autoimmune diseases requiring immunosuppressive treatment (with exceptions).
* Any form of primary or secondary immunodeficiency.
* Risk of organ perforation or bleeding as judged by the investigator.
* Severe systemic hypersensitivity reactions to study drugs/components. - Received live attenuated vaccines within 4 weeks prior to signing informed consent.
* Participated in another clinical study within 4 weeks prior to signing informed consent.
* History of another malignancy within the past 5 years, except for adequately treated non-melanoma skin cancer or in situ cancers.
* Diagnosed with neuropsychiatric disorders or any condition deemed by the investigator as unsuitable for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The safety of UCLH801 cells in patients with advanced malignant solid tumors with positive expression of CDH17 | 28 days after the CAR-T cells infusion
  The number and severity of dose-limiting toxicity (DLT) events and all adverse events occurring in subjects following the infusion of UCLH801 cells; The determination of the recommended Phase II dose (RP2D). Periodic analysis may be conducted during the dose esclation stage, including subgroup analysis, such as CDH17 expression strength, prior therapy lines and tumor burden.

SECONDARY OUTCOMES:
Evaluate the preliminary response rate of UCLH801 cells in patients with advanced malignant solid tumors expressing CDH17. | 64 days
  Efficacy: Evaluated based on objective response rate (ORR) and disease control rate (DCR)
Evaluate the pharmacodynamic (PD) characteristics of UCLH801 cells in subjects | 28 days
  Pharmacodynamics: Cytokine levels in blood/serum at various time points, including IL-2, IL-6, IL-8, IL-10, TNF-α, and IFN-γ.
Evaluate the concentration of anti-UCLH801 cell antibodies in serum | 28 days
  The production of anti-UCLH801 cell antibodies in serum
Evaluate the preliminary response rate of UCLH801 cells in patients with advanced malignant solid tumors expressing CDH17. | 2 years
  Evaluate the PFS and OS of all enrolled patients
Evaluate the peak plasma concentration (Cmax) of UCLH801 cells | 28 days
  After cell infusion, the peak concentration (Cmax), time to reach peak concentration (Tmax)
Evaluate the long-time area under the curve (AUC) of UCLH801 cells. | 90 days
  Pharmacokinetics: After cell infusion, the area under the curve (AUC) from 0 to 90 days (AUC0-90) of UCLH801 cells in peripheral blood.
Evaluate the area under the plasma concentration versus time curve (AUC) of UCLH801 cells | 28 days
  After cell infusion, evaluate the area under the curve (AUC) from 0 to 28 days (AUC0-28)

OTHER OUTCOMES:
Explore the changes in T cell infiltration and tumor microenvironment components in tumor tissues before and after UCLH801 cell infusion. | 64 days
  The distribution, quantity, and proportion of Anti-CDH17 CAR+ T cells, Treg cells, MDSCs, TAMs, TAFs, etc., in tumor tissues before and after UCLH801 cell infusion.
Explore the changes in T cell phenotype, function, persistence, and gene expression profile, and their correlation with clinical response. | 64days
  The expression and proportion of T cell surface markers (CD3, CD4, CD8, CD45RA, CD95, IL-2Rβ, CCR7, CD62L, PD1, TIM-3, LAG-3, etc.) in peripheral blood, tumor tissue, and pleural/ascitic fluid.
  Single-cell transcriptomic analysis of T cells in peripheral blood, tumor tissue, and pleural/ascitic fluid.
Subgroup evaluation of the preliminary response rate of UCLH801 cells in patients with different expressing level of CDH17. | 64 days
  Subgroup evaluation of the ORR and DCR of UCLH801 cells in patients with different expressing level of CDH17
Subgroup evaluation of the survival time of UCLH801 cells in patients with different expressing level of CDH17. | 64 days
  Subgroup evaluation of the PFS and OS of UCLH801 cells in patients with different expressing level of CDH17
Subgroup evaluation of the survival time of UCLH801 cells in patients with different tumor burden level. | 64 days
  Subgroup evaluation of the PFS and OS of UCLH801 cells in patients with different tumor burden level.
Subgroup evaluation of the preliminary response rate of UCLH801 cells in patients with different tumor burden level. | 64 days
  Subgroup evaluation of the ORR and DCR of UCLH801 cells in patients with different tumor burden level.
Subgroup evaluation of the preliminary response rate of UCLH801 cells in patients with different tumor histology. | 64 days
  Subgroup evaluation of the ORR and DCR of UCLH801 cells in patients with different tumor histology.
Subgroup evaluation of the survival time of UCLH801 cells in patients with different tumor histology. | 64 days
  Subgroup evaluation of the PFS and OS of UCLH801 cells in patients with different tumor histology.
Subgroup evaluation of the survival time of UCLH801 cells in patients with different prior therapeutic regimens. | 64 days
  Subgroup evaluation of the PFS and OS of UCLH801 cells in patients with different prior therapeutic regimens.
Subgroup evaluation of the preliminary response rate of UCLH801 cells in patients with different prior therapeutic regimens. | 64 days
  Subgroup evaluation of the ORR and DCR of UCLH801 cells in patients with different prior therapeutic regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No